CLINICAL TRIAL: NCT04019262
Title: Short Course Chemo-Radiation Therapy for Patients With Newly Diagnosed Glioblastoma: Comparison of Two Established Schedules
Brief Title: Short Course Chemo-Radiation Therapy for Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Flickinger (Other)
Responsible Party: Sponsor-Investigator, John Flickinger, Professor of Radiation Oncology & Neurosurgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 19-022
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
Keywords: Chemo-Radiation Therapy; temozolomide; lymphocytopenia
MeSH Terms: conditions — Glioblastoma; Lymphopenia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 40 Gy in 15 fractions (Active Comparator): Patients randomized to 40 Gy in 15 fractions will receive 75 mg/m^2 temozolomide per day for 15 days starting the first day of radiotherapy. This treatment will be followed by standard monthly 5 day cycles at 150 mg/m^2 for upto 1 year.
  Interventions: Radiation: Radiation Therapy; Drug: Temozolomide Oral Product
- 25 Gy in 5 fractions (Active Comparator): Patients randomized to 25 Gy in 5 fractions will receive 150 mg/m^2 temozolomide per day for 5 days starting the first day of radiotherapy. This treatment will be followed by standard monthly 5 day cycles at 150 mg/m^2 for upto 1 year.
  Interventions: Radiation: Radiation Therapy; Drug: Temozolomide Oral Product

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation
Drug: Temozolomide Oral Product — Oral Temozolomide (150mg/m^2 or 75 mg/m^2)

SUMMARY:
This is a prospective, randomized, open-label, exploratory trial of temozolomide-based chemo-radiotherapy which compares two widely used established radiation schedules with either 40 Gy in 15 fractions or 25 Gy in 5 fractions with concurrent temozolomide for both schedules in patients with glioblastoma.

DETAILED DESCRIPTION:
All patients in the study will receive usual care with short-course radiotherapy (RT) and TMZ-chemo pills.

There are three phases of treatment in this study: the Chemo-radiation Phase, the Adjuvant Phase, and the Follow-Up Phase.

Twenty-eight or fewer days prior to starting the Chemo-radiation Phase, patients will have a baseline Magnetic Resonance Imaging (MRI) scan.

Chemo-radiation Phase: In this, patient will be assigned to either a one week or a three week treatment group with radiation treatments given approximately 5 days a week as directed by the study doctor. During this time they will also take TMZ-chemo orally (by mouth) once a day on every evening including weekends starting the evening of the day that you start radiotherapy. Once radiation is completed, you will stop taking TMZ-chemo for approximately 4 weeks before going to the next phase.

Radiation therapy: Patients will be randomized between standard radiation treatment at UPMC Radiation Oncology facilities included in this protocol with either 40 Gy in 15 fractions or 25 Gy in 5 fractions, using 6 to 23 MV x-rays along with concurrent temozolomide chemotherapy for both treatment schedules.

* Clinical treatment volumes (CTV) will include all contrast enhancing tumor plus 1.7cm expansion into brain tissue (not crossing the tentorium) and all T2 FLAIR hyperintensity plus 7mm expansion into brain tissue (not crossing the tentorium). A planning target volume (PTV) expansion of 3mm will be then added to the CTV. No additional exclusion of brainstem or optic nerves is required as both treatment schedules are within tolerance.
* Treatment may be delivered with either 3D-conformal or intensity modulated radiotherapy (IMRT) techniques.

Adjuvant Phase: In the Adjuvant Phase, you will receive standard monthly 5 day cycles of TMZ-chemo at 150 mg/m^2 per day for up to 1 year.

Chemotherapy: Patient will receive concurrent temozolomide throughout radiation therapy, followed by standard monthly 5 day cycles for up to 1 year. Patients randomized to 25 Gy in 5 fractions will receive 150 mg/m^2 of temozolomide per day for 5 days starting first day of radiotherapy. Patients randomized to 40 Gy in 15 fractions will receive 75 mg/m2 of temozolomide per day for 19 days starting first day of radiotherapy. Patients will be appropriately pre-medicated with anti-nausea medication, prior to taking temozolomide. All patients will also receive prophylactic treatment for pneumocystis pneumonia with Bactrim or other alternative antibiotics if allergic.

Follow-up Interval: Procedures performed to evaluate the safety and effectiveness of the study procedures are called "monitoring" or "follow-up" procedures. Subject participants will not be scheduled for any additional follow-up visits for this study than they would normally have if they were not in this study. Radiation Oncologists and Neuro-Oncologists usually see their patients one month after the first chemo-radiotherapy cycle before starting the next cycle of chemotherapy. After that Neuro-Oncologists and Radiation Oncologists will see the patients every 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria for study enrollment:

* Age ≥18 with ability to provide written informed consent
* Pathologically confirmed WHO Grade IV Gliobastoma prior receiving radiotherapy
* Prior radiotherapy to a dose of ≥50Gy
* No signs of distant metastases
* Baseline laboratory assessment including CBC and blood chemistry, ANC > or equal 1500, Platelet count greater or equal 100. Liver function tests and creatinine not greater than twice ULN.
* Patient should not be pregnant. Urine or blood β-HCG within 14 days prior to study start for females who are not atleast one year post-menopausal or who have ot undergone a surgical sterilization procedure
* A baseline MRI scan of the brain is required to determine how much tumor is present for properly planning patient's radiotherapy.
* Karnofsky Performance Status (KPS) below 60 or ECOG of 3 or 4
* Any number or type of prior chemotherapy is allowed (patient may receive concurrent or adjuvant systemic therapy such as cetuximab at the discretion of the treating oncologic team).

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible for enrollment:

* Evidence of distant metastases on any staging or imaging modality
* Women who are breast feeding, or have a positive pregnancy test (reproductive age should use effective birth control during study)
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the principal investigator.
* Karnofsky Performance Status less than 50
* Prior radiotherapy to involved site in brain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 9 years
  The length of time from the start of treatment that patients remain alive.
Change in Absolute Lymphocyte Count | From baseline up to 5 years.
  Differences in absolute lymphocyte count (total lymphocyte count <800 - 500/mm^3 <0.8 - 0.5 x 10^9 /L) / total # patients, during treatment.

SECONDARY OUTCOMES:
Progression free survival (PFS) - 25 Gy in 5 fractions | Up to 9 years
  The length of time during and after the treatment that a patient lives without worsening disease per Response Assessment in Neuro-Oncology (RANO) criteria. Disease progression per RANO: (any of the following): ≥25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids*; significant increase in T2/FLAIR nonenhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy* not caused by comorbid events; any new lesion; clear clinical deterioration not attributable to other causes apart from the tumor (eg, seizures, medication adverse effects) or changes in corticosteroid dose; failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease.
Progression free survival (PFS) - 40 Gy in 15 fractions | Up to 9 years
  The length of time during and after the treatment that a patient lives without worsening disease per Response Assessment in Neuro-Oncology (RANO) criteria. Disease progression per RANO: (any of the following): ≥25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids*; significant increase in T2/FLAIR nonenhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy* not caused by comorbid events; any new lesion; clear clinical deterioration not attributable to other causes apart from the tumor (eg, seizures, medication adverse effects) or changes in corticosteroid dose; failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease.

CONTACTS AND LOCATIONS:
Overall Officials: John Flickinger, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No